CLINICAL TRIAL: NCT05563636
Title: Efficacy of High Voltage VS Standard Voltage Radiofrequency on Unilateral Lower Limb Neuralgia in a Patient With Failed Back Surgery Syndrome
Brief Title: High Voltage VS Standard Voltage Radiofrequency in a Patient With Failed Back Surgery Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amani Hassan Abdel-Wahab, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AssiutU_HAA_RFA
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Neuralgia; Failed Back Surgery Syndrome
MeSH Terms: conditions — Neuralgia; Failed Back Surgery Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (group S) (Other): patients will be given standard PRF treatment: temperature 42 ℃, frequency 2 Hz, pulse width 20 ms, voltage 37-41 V, time 120 s.
  Interventions: Device: standard pulsed radio frequency (PRF)
- group H (Experimental): patients will be given high-voltage long-term PRF treatment: temperature 42 ℃, frequency 2 Hz, pulse width 20 ms, the voltage range of 50-90 V, At the beginning, the patient will feel a severe burning sensation in the original pain area, and slowly after the patient tolerates it. Increase the voltage and gradually increase to the maximum voltage that the patient can tolerate (up to 70-90 V) until the end of 900 s.
  Interventions: Device: high-voltage long-term pulsed radio frequency (PRF)

INTERVENTIONS:
Device: standard pulsed radio frequency (PRF) — patients will be given standard pulsed radiofrequency (PRF) treatment: temperature 42 ℃, frequency 2 Hz, pulse width 20 ms, voltage 37-41 V, time 120 s.
  Other Names: control group
  Arms: control (group S)
Device: high-voltage long-term pulsed radio frequency (PRF) — patients will be given standard pulsed radiofrequency (PRF) treatment: temperature 42 ℃, frequency 2 Hz, pulse width 20 ms, voltage 50-90 V, At the beginning, the patient will feel a severe burning sensation in the original pain area, and slowly after the patient tolerates it. Increase the voltage and gradually increase to the maximum voltage that the patient can tolerate (up to 70-90 V) until the end of 900 s.
  Arms: group H

SUMMARY:
Postoperative lumbar spine pain syndrome (FBSS) refers to patients who have undergone surgery for lumbar spine disease one or more times and still have intractable lumbosacral pain after surgery, with or without lower limb sensory and motor dysfunction. Pain is the main reason for reducing patients' quality of life. Hussain and Erdek believe that despite up to 3 months of postoperative intervention, pain may still exist. Since persistent pain seriously affects patients' daily life and work, optimizing the FBSS treatment plan and improving the quality of life of FBSS patients cannot be ignored. At present, the treatment methods for neuropathic pain radiated to the lower extremity after lumbar spine surgery mainly include oral drug therapy, nerve block, pulsed radio frequency (PRF) and spinal cord electrical stimulation, and other minimally invasive interventional methods. Still, there is no domestic or foreign treatment method is reported in the literature to be effective.

DETAILED DESCRIPTION:
Selective nerve root PRF is an effective method for treating neuropathic pain, but its analgesic mechanism is still unclear. The traditional PRF adopts the standard 42 ℃ mode, but due to its low voltage (40 V), short duration (120 s), and limited intensity of action, the patient cannot get the best therapeutic effect. In recent years, high-voltage long-term PRF has been gradually applied to treating neuropathic pain such as postherpetic neuralgia, trigeminal neuralgia, and glossopharyngeal neuralgia, and achieved ideal results.

. Selective spinal nerve puncture under ultrasound and X-ray guidance: After the patient enters the operating room, the venous access is inserted, and the patient is placed in a prone position. ECG monitoring is given, and the patient's vital signs are continuously monitored. Routine sterilization and laying of sheets, puncture with an 20 G radiofrequency puncture needle under the guidance of ultrasound, repeated X-rays to confirm the position of the needle tip, when the needle tip reaches the target position, the X-ray front view will show that the needle tip of the puncture needle is located below the pedicle, and the lateral view shows The tip of the puncture needle is located at the posterior 1/2of the intervertebral foramen, then connect the radiofrequency treatment apparatus, perform sensory and motor tests, and perform sensory tests The pain in the corresponding innervated area is reproduced within 0.5 V and 50 Hz, and is consistent with the patient's original pain location; if >0.5 V does not induce pain in the original pain area, fine-tune the needle tip position and then perform the sensory test until 0.1 The needle tip position can be fixed when the patient's original pain can be induced within ~0.5 V. In the exercise test, muscle beats in the corresponding area were induced within 1.0 V and 2 Hz. After the test was successful, 1 ml of contrast agent will be injected, and the X-ray should show that the contrast agent spread along the nerve root and epidural space.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a history of lumbar spine surgery without instrumentation. , have clear symptoms of lumbar nerve root irritation, and unilateral lower extremity symptoms, and the straight leg raising test is positive

Exclusion Criteria:

* Mechanical compression to nerve root
* Spondylolisthesis, retrolithesis
* Spondylodiscitis
* Lumbar canal stenosis
* Inflammatory low back pain
* Coagulopathy
* Local anesthetic allergy
* Infection at the site of injection
* Systemic infection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
change in Oswestry Disability Index (ODI) | assessing a change in Change ODI from Baseline at 6 months
  assessing a change in Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: Amani H Abdel-wahab, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No